CLINICAL TRIAL: NCT05258006
Title: Clinical and Radiographic Assessment of Autogenous Dentin Nanoparticles in Treatment of Stage III Periodontitis: A Split-Mouth Clinical Study
Brief Title: Assessment of Autogenous Dentin Graft in Treatment of Infra-bony Defect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Professor of Periodontology, October 6 University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2022-02-10; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Periodontitis (Stage 3)
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open flap debridement + allograft bone (Maxgraft) (Placebo Comparator)
  Interventions: Procedure: Autogenous demineralized dentin nanoparticles
- Open flap debridement + Autogenous demineralized nanoparticles (Active Comparator)
  Interventions: Procedure: Autogenous demineralized dentin nanoparticles

INTERVENTIONS:
Procedure: Autogenous demineralized dentin nanoparticles — Effect of Autogenous demineralized dentin nanoparticles in bone gain in infrabony defect

SUMMARY:
The aim of the present study was to evaluate the effect of demineralized autogenous dentine on treatment of infrabony defects.

DETAILED DESCRIPTION:
In this study, the investigators tested the effect of demineralized autogenous dentine as a bone graft in treatment of stage III periodontitis in term of probing pocket depth reduction, mean gain in clinical attachment level, and bone gain in defect sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good systemic health and no contraindication for periodontal surgery.
* Patients who are able to maintain good oral hygiene.
* Gingival thickness for the site selected should be ≥1mm.
* Probing depth of ≥ 6mm.
* Patient has at least one hopeless teeth

Exclusion Criteria:

* Active infectious diseases (hepatitis, tubercu¬losis, HIV, etc….).
* Medically compromised patients.
* Smokers and alcoholic abusers
* People who suffer from any systemic disease that affect the periodontium.
* Pregnant, postmenopausal women.
* People who take anti-inflammatory drugs, anti¬biotics or vitamins within the previous 3 month.
* People who use mouth washes regularly
* Participants in other clinical trials.

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Vertical bone loss | 6 months
  vertical bone loss was measured from cementoenamel junction (CEJ) to the base of the bone defect in each site in group I & II.
Clinical attachment level | 6 months
  Clinical attachment level was measured at baseline and 6 months
Probing pocket depth | 6 months
  Probing pocket depth was measured at baseline and 6 months
Bone gain | 6 months
  The bone gain is calculated by:
  * Preoperative VBL (at baseline): measured as the distance from cementoenamel junction (CEJ) to the base of the bone defect.
  * Postoperative VBL (after 6 months) measured as the distance from cementoenamel junction (CEJ) to the base of the bone formation.
  * Postoperative bone fill (bone gain after 6 months) [measured by subtracting the preoperative VBL from the postoperative VBL].

SECONDARY OUTCOMES:
Plaque Index | 6 months
  plaque index was measured at baseline, 3, 6 months
Gingival index | 6 months
  Gingival index was measured at baseline, 3, 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elgendy EA, Elgendy AM, ElBorady OM. Clinical And Radiographic Assessment Of Autogenous Dentin Nanoparticles In Treatment Of Stage Iii Periodontitis: A Split-Mouth Clinical Study. J Pak Med Assoc. 2023 Apr;73(Suppl 4)(4):S310-S316. doi: 10.47391/JPMA.EGY-S4-60. PMID 37482878